CLINICAL TRIAL: NCT07407088
Title: Effect of Virtual Reality-Supported Task-Oriented Training in Individuals With Rotator Cuff Lesions: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet CANLI, Asst. Prof., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43834581758'
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Rotator Cuff Lesions
Keywords: Rotator cuff lesions; virtual reality; task-oriented training

STUDY DESIGN:
Intervention Model Description: randomized controlled trials
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Participants allocated to the control group will receive conventional physiotherapy consisting of therapeutic exercises and electrophysical agents. The treatment program will be administered three times per week for six weeks, for a total of 18 sessions. Therapeutic exercises will focus on improving shoulder mobility, strength, and functional use of the upper extremity. Electrophysical agents will be applied as part of standard clinical practice to support pain management and tissue healing. No virtual reality-supported training will be provided to participants in this group.
  Interventions: Other: Conventional treatment
- Virtual Reality-Supported Task-Oriented Training Group (Experimental): Participants allocated to the intervention group will receive virtual reality-supported task-oriented training in addition to conventional physiotherapy. Conventional physiotherapy will consist of therapeutic exercises and electrophysical agents and will be administered three times per week for six weeks, totaling 18 sessions. The virtual reality-supported task-oriented training will be delivered during the same treatment period and will include functional, goal-directed activities simulating activities of daily living, such as kitchen-related tasks, cleaning activities, and pushing and pulling movements.
  The virtual reality program will be performed using a virtual reality device and will be tailored to the participant's functional capacity and tolerance, with task difficulty progressively adjusted throughout the intervention period. The training aims to enhance shoulder function, upper extremity use, motor performance, and psychosocial outcomes by promoting active participation and
  Interventions: Other: Conventional treatment; Other: Virtual Reality-Supported Task-Oriented Training

INTERVENTIONS:
Other: Conventional treatment — The treatment program will be administered three times per week for six weeks, for a total of 18 sessions. Therapeutic exercises will focus on improving shoulder mobility, strength, and functional use of the upper extremity. Electrophysical agents will be applied as part of standard clinical practice to support pain management and tissue healing.
Other: Virtual Reality-Supported Task-Oriented Training — he virtual reality-supported task-oriented training will be delivered during the same treatment period and will include functional, goal-directed activities simulating activities of daily living, such as kitchen-related tasks, cleaning activities, and pushing and pulling movements.
  The virtual reality program will be performed using a virtual reality device and will be tailored to the participant's functional capacity and tolerance, with task difficulty progressively adjusted throughout the intervention period. The training aims to enhance shoulder function, upper extremity use, motor performance, and psychosocial outcomes by promoting active participation and graded exposure to functional movements.
  Arms: Virtual Reality-Supported Task-Oriented Training Group

SUMMARY:
Rotator cuff lesions are among the most common causes of shoulder pain and functional limitation, often affecting daily living activities and quality of life. Conventional physiotherapy interventions such as therapeutic exercises and electrophysical agents are widely used; however, persistent pain, kinesiophobia, and functional disability may limit treatment outcomes. Virtual reality-supported task-oriented training has emerged as a promising rehabilitation approach by providing immersive, functional, and goal-directed activities that may enhance motor performance and psychosocial outcomes.

The aim of this randomized controlled trial is to investigate the effects of virtual reality-supported task-oriented training added to conventional physiotherapy in individuals with rotator cuff lesions. Participants will be randomly allocated into two groups: a control group receiving conventional physiotherapy (therapeutic exercises and electrophysical agents) and an intervention group receiving virtual reality-supported task-oriented training in addition to conventional physiotherapy. Both groups will undergo treatment three times per week for six weeks, totaling 18 sessions.

Outcome measures will include pain intensity at rest, during activity, and at night assessed by the Visual Analog Scale (VAS); grip strength measured by dynamometry; pinch strength measured by pinchmeter; upper extremity function assessed using the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire; shoulder pain and disability assessed by the Shoulder Pain and Disability Index (SPADI); kinesiophobia assessed by the Tampa Scale of Kinesiophobia; pain catastrophizing assessed by the Pain Catastrophizing Scale; and anxiety and depression assessed using the Hospital Anxiety and Depression Scale (HADS). The findings of this study are expected to contribute to evidence-based rehabilitation strategies for individuals with rotator cuff lesions.

DETAILED DESCRIPTION:
Rotator cuff lesions are a leading cause of shoulder pain, reduced range of motion, muscle weakness, and functional limitations, significantly affecting activities of daily living. In addition to physical impairments, individuals with rotator cuff lesions often experience psychosocial factors such as kinesiophobia, pain catastrophizing, anxiety, and depression, which may negatively influence rehabilitation outcomes. Conventional physiotherapy interventions, including therapeutic exercises and electrophysical agents, are commonly prescribed; however, these approaches may not adequately address functional task performance and psychosocial components of recovery.

Task-oriented training focuses on practicing meaningful, goal-directed activities that closely resemble real-life tasks, thereby facilitating motor learning and functional improvement. Recently, virtual reality-supported rehabilitation has gained increasing attention as it enables the simulation of functional environments, provides multisensory feedback, and enhances patient engagement and motivation. Virtual reality-supported task-oriented training may offer additional benefits by integrating physical and cognitive demands while reducing fear of movement through graded exposure to functional tasks.

This randomized controlled trial aims to investigate the effectiveness of virtual reality-supported task-oriented training when added to conventional physiotherapy in individuals with rotator cuff lesions. Eligible participants will be randomly assigned to either a control group or an intervention group using a random allocation method. The control group will receive conventional physiotherapy consisting of therapeutic exercises and electrophysical agents. The intervention group will receive the same conventional physiotherapy program plus virtual reality-supported task-oriented training. Both interventions will be administered three times per week for six weeks, resulting in a total of 18 treatment sessions.

The virtual reality-supported task-oriented training program will include functional tasks designed to simulate activities of daily living, such as kitchen-related activities, cleaning tasks, and pushing and pulling movements. These tasks will be performed using a virtual reality device and will be progressively adapted according to the participant's functional level and tolerance. The training is intended to promote upper extremity use, improve shoulder function, and address psychosocial factors associated with pain and movement avoidance.

Assessments will be conducted before and after the intervention period. Pain intensity at rest, during activity, and at night will be evaluated using the Visual Analog Scale (VAS). Grip strength of the affected side will be measured using a hand dynamometer, and pinch strength will be assessed using a pinchmeter. Upper extremity functional status will be evaluated using the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, while shoulder-specific pain and disability will be assessed using the Shoulder Pain and Disability Index (SPADI). Kinesiophobia will be measured using the Tampa Scale of Kinesiophobia, pain catastrophizing using the Pain Catastrophizing Scale, and psychological status using the Hospital Anxiety and Depression Scale (HADS).

The results of this study will provide evidence regarding the effectiveness of virtual reality-supported task-oriented training as an adjunct to conventional physiotherapy in improving pain, strength, functional outcomes, and psychosocial factors in individuals with rotator cuff lesions. The findings may help guide clinical decision-making and the development of innovative, functionally oriented rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Diagnosed with a rotator cuff lesion confirmed by clinical examination and/or imaging methods (MRI or ultrasound)
* Presence of shoulder pain and functional limitation for at least 3 months
* Ability to actively use the affected upper extremity
* Ability to understand and follow verbal instructions
* Willingness to participate in the study and provide written informed consent

Exclusion Criteria:

* History of shoulder surgery on the affected side
* Full-thickness rotator cuff tear requiring surgical intervention
* Presence of shoulder fracture, dislocation, or acute traumatic injury within the last 6 months
* Neurological disorders affecting the upper extremity (e.g., stroke, multiple sclerosis, peripheral neuropathy)
* Systemic inflammatory or rheumatologic diseases affecting the shoulder (e.g., rheumatoid arthritis)
* Severe cervical spine pathology with referred shoulder pain
* Severe visual, vestibular, or cognitive impairments that may limit participation in virtual reality training
* Current participation in another structured shoulder rehabilitation program
* Contraindications to physical therapy or virtual reality-based interventions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Upper extremity functionality | 6 week
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will be used to assess upper extremity functional disability. The DASH is a self-reported outcome measure consisting of 30 items that evaluate difficulty in performing physical activities and the severity of symptoms related to upper extremity disorders. Scores range from 0 to 100, with higher scores indicating greater disability.

SECONDARY OUTCOMES:
Pain Intensity (Visual Analog Scale - VAS) | 6 week
  Pain intensity at rest, during activity, and at night will be assessed using the Visual Analog Scale (VAS). The VAS consists of a 10-cm horizontal line representing pain intensity, where 0 indicates "no pain" and 10 indicates "worst imaginable pain."
Grip Strength | 6 week
  Grip strength of the affected upper extremity will be measured using a hand dynamometer. Measurements will be recorded in kilograms, and higher values indicate greater grip strength.
Pinch Strength | 6 week
  Pinch strength of the affected upper extremity will be assessed using a pinchmeter. Measurements will be recorded in kilograms, with higher values indicating greater pinch strength.
Disability | 6 week
  The Shoulder Pain and Disability Index (SPADI) will be used to assess shoulder-related pain and functional disability. The questionnaire consists of pain and disability subscales, with total scores ranging from 0 to 100; higher scores indicate greater pain and disability.
Kinesiophobia | 6 week
  Kinesiophobia will be evaluated using the Tampa Scale of Kinesiophobia, which measures fear of movement and re-injury related to pain. Higher scores indicate greater levels of kinesiophobia.
Pain Catastrophizing | 6 week
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale, which evaluates exaggerated negative cognitive and emotional responses to pain. Higher scores reflect greater pain catastrophizing.
Anxiety and Depression | 6 week
  Psychological status will be assessed using the Hospital Anxiety and Depression Scale (HADS), which consists of anxiety and depression subscales. Higher scores indicate greater levels of anxiety and depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet CANLI, Ph.D., Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No